CLINICAL TRIAL: NCT03957902
Title: Assessment of Direct Biomarkers of Aspirin Action to Develop a Precision Chemoprevention Therapy of Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); G. d'Annunzio University (Other); Hospital Clínico Universitario Lozano Blesa (Other)
Responsible Party: Principal Investigator, Ángel Lanas Arbeloa, Head of Digestive Diseases Service, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PI17/01109; 2018-002101-65 (EudraCT Number)
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (100 mg/24h) (Experimental)
  Interventions: Drug: acetylsalicylic acid
- Arm 2 (300 mg/24h) (Experimental)
  Interventions: Drug: acetylsalicylic acid
- Arm 3 (100 mg/12h) (Experimental)
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: acetylsalicylic acid — Different dosage effect over platelet COX enzymes, non- neoplastic and neoplastic colonic tissues used as biomarkers of clinical efficacy in CRC chemoprevention

SUMMARY:
Acetylsalicylic acid (ASA) seems the ideal colorectal cancer (CRC) chemoprevention agent. Several ongoing trials are testing the effect of ASA as co-therapy in CRC. The mechanisms of action, the appropriate dose and the ideal target population are unknown. The investigators have demonstrated that doses of 100 mg of ASA induce direct and partial but persistent acetylation of the cyclooxygenase (COX) isoenzyme COX-1 in the normal colorectal mucosa. The primary objective is to perform a study of aspirin by using a proteomic assay for comparing platelet COX-1 and CRC mucosal COX-1 after different doses of ASA. Secondary objectives are: the measurement of prostaglandin E2 (PGE2) and phosphorylated S6 protein (p-S6) levels in CRC mucosa, the assessment of indirect biomarker of aspirin action (serum thromboxane B2 (TXB2) and urinary levels of 11-dehydro-TXB2 (TX-M)), the evaluation of systemic biomarkers of inflammatory/tumorigenic COX-2 by assessing urinary levels of major metabolite of PGE2 (PGE-M). Methods: Phase II randomized clinical trial in 60 patients with newly diagnosed CRC in 3 groups of 20 patients receiving 100 or 300 mg/day, or 100 mg/12 hours of enteric-coated ASA for 3±1 weeks, prior to definitive treatment by surgery. Main outcome: Acetylation of COX-1 and COX-2. Eicosanoid levels in target organs. Expected results: Evidence for the current uncertainty about the mechanisms of action and the dose required to obtain the best chemopreventive effect with ASA in CRC. Confirm acetylation of COX as a key biomarker of efficacy with ASA.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 < 80 years old
* recent diagnosis (< 48h) of rectum or colon cancer, established by endoscopy and later confirmed by anatomo-pathologic study
* normal coagulation values and biochemical vales without clinically significant deviations that, at the discretion of the investigator, may interfere with the study procedures

Exclusion Criteria:

* Allergy to ASA or to any other NSAID.
* Rectal cancer requiring neoadjuvant treatment within the two weeks following the beginning of ASA treatment.
* Previous use of ASA, NSAIDs, antiplatelet agents, corticosteroids or misoprostol within the 15 days prior to diagnosis and/or anticipation of need for treatment with any of these drugs during the study period. History of peptic ulcer disease or active peptic ulcer or any other gastrointestinal disease that may be considered a contraindication to the use of ASA, without the concomitant use of proton pump inhibitors.
* Diagnosis of bleeding disorders.
* Diagnosis of cancer (excluding non-melanoma skin cancer) within the previous 3 years.
* Conditions supposing serious comorbidity, excluding diabetes, and including respiratory, cardiac, hepatic and renal diseases.
* Active smoking.
* Pregnancy or breastfeeding.
* History of drug or alcohol abuse.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in acetylation levels of COX enzymes in platelets and non-neoplastic and neoplastic colonic tissues | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment

SECONDARY OUTCOMES:
Assessment of changes in prostaglandin E2 (PGE2) levels in colorectal mucosa depending on drug dosis | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment
Assessment of changes in phosphorylated S6 protein (p-S6) levels in colorectal mucosa depending on drug dosis | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment
Assessment of changes in thromboxane B2 (TxB2) levels in urine as indirect systemic biomarker depending on drug dosis | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment
Assessment of changes in urinary metabolite 11-dehydro-TxB2 (TX-M) levels as indirect systemic biomarker depending on drug dosis | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment
Assessment of changes in major urinary metabolite of PGE2 (PEG-M) levels depending on drug dosis | before the beginning of the treatment and 3 ± 1 weeks of acetylsalicylic acid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Lanas Arbeloa, MD, Principal Investigator — Instituto de Investigación Sanitaria Aragón
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patrignani P, Tacconelli S, Contursi A, Piazuelo E, Bruno A, Nobili S, Mazzei M, Milillo C, Hofling U, Hijos-Mallada G, Sostres C, Lanas A. Optimizing aspirin dose for colorectal cancer patients through deep phenotyping using novel biomarkers of drug action. Front Pharmacol. 2024 Feb 29;15:1362217. doi: 10.3389/fphar.2024.1362217. eCollection 2024. PMID 38495101